CLINICAL TRIAL: NCT01834820
Title: Pilot Study: Epinephrine, Dexamethasone, and Hypertonic Saline in Children With Bronchiolitis, Randomised Clinical Trial of Efficacy and Safety
Brief Title: Epinephrine, Dexamethasone, and Hypertonic Saline in Bronchiolitis, Randomised Clinical Trial of Efficacy and Safety
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital General Naval de Alta Especialidad - Escuela Medico Naval (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: HGNAE-01
Record Dates: First submitted 2013-01-15; First posted 2013-04-18 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; Epinephrine; Dexamethasone; Hospitalization; Hypertonic Saline
MeSH Terms: conditions — Bronchiolitis | interventions — Epinephrine; Dexamethasone; Saline Solution, Hypertonic; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Epinephrine and Dexamethasone (Experimental): First day: One treatment of nebulized dexamethasone 4mg (1ml of dexamethasone 8mg/2ml) + 3ml NS, followed by two treatments of nebulized epinephrine (3 ml of epinephrine in a 1:1000 solution per treatment) with interval 20 minutes. And one treatment of nebulized dexamethasone every 24h for three days.
  Interventions: Drug: Epinephrine and Dexamethasone
- Hypertonic Saline 3% (Experimental): 3 treatments of nebulized HS 3% 4ml in first day of treatment with interval 20 minutes And one treatment of nebulized HS 3% 4ml every 24 hours for 3 days
  Interventions: Drug: Hypertonic Saline
- Normal Saline 0.9% (Active Comparator): 3 treatments of nebulized Normal Saline 0.9% 4ml in first day of treatment with interval 20 minutes. And one treatment of nebulized Normal Saline 0.9% 4ml every 24 hours for 3 days
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Epinephrine and Dexamethasone
  Arms: Epinephrine and Dexamethasone
Drug: Hypertonic Saline
  Arms: Hypertonic Saline 3%
Drug: Normal Saline
  Arms: Normal Saline 0.9%

SUMMARY:
In infancy, bronchiolitis is the most common acute infection of the lower respiratory Tract. The current treatment of bronchiolitis is controversial. Bronchodilators and corticosteroids are widely used but not routinely recommended. Hypertonic saline is currently the only drug recommended by the Spanish Association of Pediatrics in treatment guidelines.

The purpose of this study is quantify whether epinephrine, dexamethasone, and hypertonic saline are effective to decrease the rate of hospital admissions at seven day, also verify adverse effects in patients submitted.

DETAILED DESCRIPTION:
Infections remain the leading cause of death globally, in 2010 from 7.6 million deaths in children under 5 years, 64% is attributed to an infectious cause, acute lower respiratory tract include 14.1% of all deaths, representing the leading cause of global mortality in children. In Mexico in children under 15 years the leading cause of death are conditions originating in the perinatal period, congenital malformations deformities and chromosomal abnormalities and third lower airway infections.

Bronchiolitis being the leading cause of lower respiratory tract infection in infants, with a global load elevated, represented by a hospitalization rate of 3% of the total population of children under one year. Estimated that only in the United States of America, the annual cost of hospitalizations of patients under one year with bronchiolitis exceeds $ 700 million / year. Unfortunately, there is evidence that hospital admission rates have increased almost twice in the last 10-15 years in the United States and Canada, and it occurs most impact in developing countries, where befall 99% of deaths related to Respiratory Syncytial Virus (RSV), the leading cause of infection of lower airways.

The etiology of the disease is attributed by 50 to 80% of all cases the RSV worldwide, has been reported in Mexico RSV as a cause of just over 80% of infections lower airway requiring hospitalization.

Given such alarming morbidity figures, note that the mortality from this disease is low, representing less than 400 deaths annually, perhaps explained by the wide clinical spectrum that presents.

Currently no management guide recommends specific treatment for bronchiolitis, in particular, it is necessary to mention the national clinical practice guideline, which emphasizes that there is no consensus on proper drug treatment for this disease.

Until 2006, the American Academic of Pediatrics guidelines and Scottish Intercollegiate Guidelines Network recommend not using any systemic or inhaled drug for the management of bronchiolitis, this widely shown including bronchodilators, corticosteroids, antivirals and antitussive.

Recent review of Cochrane Acute Respiratory Infections Group about benefit of glucocorticoids for acute viral bronchiolitis, concluded not significantly reduce outpatient admissions by days 1 and 7 when compared to placebo and there was no benefit in length of stay for inpatients; however unadjusted results from a large factorial low risk o bias Randomized Controlled Trial found combined high-dose systemic dexamethasone and inhaled epinephrine reduced admissions 26% with no differences in short-term adverse effects.

L. Hartling et al, in 2011 review demonstrates the superiority of epinephrine compared to placebo for short-term outcomes for outpatients, particularly in the first 24 hours of care.

In Mexico there is evidence of the use of dexamethasone in combination with inhaled salbutamol in the management of patients with bronchiolitis with decreased hospital stay to 24hrs 96% vs 75% at P <0.05

Furthermore, hypertonic saline (HS) has proven effective with minimal adverse effects and thus, currently the clinical practice guidelines of Spain in 2010, are the only recommended method.

A study conducted by Ipek et al, a comparative study with four treatment groups I Salbutamol + Normal Saline 0.9% (NS), Group II Salbutamol + HS, Group III HS and Group IV NS, with the measurement variables heart rate, respiratory difficulty scale, and oxygen saturation, found that after treatment in all groups were significant improvement in breathlessness p <0.0001. These findings demonstrate the self-limiting nature of disease, bringing the ethical basis using NS as a control group because, per se, significantly reduces respiratory distress and as indicated by the clinical practice guidelines as part of management symptomatic.

Therefore this research aims to be a pilot study to the population of Marina, first, get the best treatment evidence, using treatments that have reported better results in order to establish optimal treatment to reduce the rate of hospital admissions and with minimal adverse effects.

Included in the study, patients with mild to moderate bronchiolitis, defining it as the first event of wheezing in infants under two years with a history of viral infection prodrome attending the emergency department (ED) the period January to April in 2013.

Supportive care including oxygen supplementation if oxygen saturation less than 92% while breathing ambient; aspiration, temperature control and hydration when necessary were provided to all patients. Infants 2 to 24 months of age with bronchiolitis who were seen at emergency department were eligible for the study if they had a score of 2 to 8 on the Clinical Bronchiolitis Severity Scores (CBSS). The CBSS values the respiratory distress with respiratory rate, wheezing, general condition and presence of retractions on a scale from 0 to 12, with higher scores indicating more severe illness; an a score above 9 very severe illness.

All eligible patients were randomly assigned to one of three groups according to the consecutive order of their admission to the ED: group I received first day one treatment of nebulized dexamethasone and two treatments of epinephrine, followed by three days one treatment nebulized dexamethasone; Group II the first day received three nebulized HS followed by treatment with HS every 24 hours for 3 days and group 3 received only NS first day 3 treatments followed one treatment every 24hrs for 3 days. The nebulized solution was administered in a double-blind setting every 20 min until 3 doses had been administered (0, 20 and 40th min).

The research recorded the patient's CBSS score, respiratory rate, heart rate, and oxygen saturation in ambient air at baseline, between the three nebulizations, and at 60 and 90 minutes; rectal temperature at baseline and 90 minutes; blood pressure at baseline and 90 minutes; and any side effects throughout the observation period in the emergency department.

Followed up each patient to record the admission rate in each group at 7 days of the study, as measure of efficacy of treatment. Likewise measured the potential adverse effects of each group, including hypertension, bronchospasm, tachycardia and any eventuality, as a security measure

ELIGIBILITY:
Inclusion Criteria:

* Patients under 2 years of age diagnosed with bronchiolitis
* Be beneficiaries Marine
* Outpatient
* Severity of Bronchiolitis mild to moderate scale according to Wood-Downes

Exclusion Criteria:

* Patients with a history of atopy
* Patients with a history of asthma in infants
* Patients with serious bacterial illness criteria
* Patients with comorbidity

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Rate of hospital admissions at seven day in infants whit bronchiolitis. | From date of randomization until the day seven of treatment
  Tracking each patient until 7 days after treatment to verify hospitalization rate

SECONDARY OUTCOMES:
Number of participants with adverse events in each arm of treatment | From date of randomization until the seven day of treatment

OTHER OUTCOMES:
Change from baseline CBSS after three treatments in the first day | First day of treatment
  Each patient on admission to the emergency department with a diagnosis of mild to moderate bronchiolitis were taken CBSS baseline, then at 20 minutes after completion three nebulized treatment in the first day.
Change from baseline heart rate after three treatments in the first day | First day of treatment
  Each patient on admission to the emergency department with a diagnosis of mild to moderate bronchiolitis were taken heart rate, then at 20 minutes after completion three nebulized treatment in the first day.
Change from baseline oxygen saturation after three treatments in the first day | First day of treatment
  Each patient on admission to the emergency department with a diagnosis of mild to moderate bronchiolitis were taken oxygen saturation, then at 20 minutes after completion three nebulized treatment in the first day.

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Rodríguez Cuevas, pediatrician, Principal Investigator
Locations (1):
- Hospital General Naval de Alta Especialidad, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Turner T, Wilkinson F, Harris C, Mazza D; Health for Kids Guideline Development Group. Evidence based guideline for the management of bronchiolitis. Aust Fam Physician. 2008 Jun;37(6 Spec No):6-13. PMID 19142264
- [Background] American Academy of Pediatrics Subcommittee on Diagnosis and Management of Bronchiolitis. Diagnosis and management of bronchiolitis. Pediatrics. 2006 Oct;118(4):1774-93. doi: 10.1542/peds.2006-2223. PMID 17015575
- [Background] Plint AC, Johnson DW, Patel H, Wiebe N, Correll R, Brant R, Mitton C, Gouin S, Bhatt M, Joubert G, Black KJ, Turner T, Whitehouse S, Klassen TP; Pediatric Emergency Research Canada (PERC). Epinephrine and dexamethasone in children with bronchiolitis. N Engl J Med. 2009 May 14;360(20):2079-89. doi: 10.1056/NEJMoa0900544. PMID 19439742
- [Background] Nair H, Nokes DJ, Gessner BD, Dherani M, Madhi SA, Singleton RJ, O'Brien KL, Roca A, Wright PF, Bruce N, Chandran A, Theodoratou E, Sutanto A, Sedyaningsih ER, Ngama M, Munywoki PK, Kartasasmita C, Simoes EA, Rudan I, Weber MW, Campbell H. Global burden of acute lower respiratory infections due to respiratory syncytial virus in young children: a systematic review and meta-analysis. Lancet. 2010 May 1;375(9725):1545-55. doi: 10.1016/S0140-6736(10)60206-1. PMID 20399493
- [Background] Zorc JJ, Hall CB. Bronchiolitis: recent evidence on diagnosis and management. Pediatrics. 2010 Feb;125(2):342-9. doi: 10.1542/peds.2009-2092. Epub 2010 Jan 25. PMID 20100768
- [Background] Noyola DE, Rodriguez-Moreno G, Sanchez-Alvarado J, Martinez-Wagner R, Ochoa-Zavala JR. Viral etiology of lower respiratory tract infections in hospitalized children in Mexico. Pediatr Infect Dis J. 2004 Feb;23(2):118-23. doi: 10.1097/01.inf.0000110269.46528.a5. PMID 14872176
- [Background] Intercollegiate S, Network G. Bronchiolitis in children. (SIGN Guideline No 91). 2006;(november).
- [Background] Nebot MS, Teruel GC, Cubells CL, Sabadell MD, Fernandez JP. [Acute bronchiolitis clinical practice guideline: recommendations for clinical practice]. An Pediatr (Barc). 2010 Oct;73(4):208.e1-10. doi: 10.1016/j.anpedi.2010.04.015. Epub 2010 Jul 14. Spanish. PMID 20634158
- [Background] Acosta A et all. Diagnóstico y manejo en niños con Bronquiolitis en fase aguda, México: Secretaria de Salud. Catálogo maestro de Guías de práctica clínica: IMSS -032-08. 2010
- [Background] Hartling L, Bialy LM, Vandermeer B, Tjosvold L, Johnson DW, Plint AC, Klassen TP, Patel H, Fernandes RM. Epinephrine for bronchiolitis. Cochrane Database Syst Rev. 2011 Jun 15;(6):CD003123. doi: 10.1002/14651858.CD003123.pub3. PMID 21678340
- [Background] Patel H, Platt R, Lozano JM. WITHDRAWN: Glucocorticoids for acute viral bronchiolitis in infants and young children. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD004878. doi: 10.1002/14651858.CD004878.pub2. PMID 18254063
- [Background] Koehoorn M, Karr CJ, Demers PA, Lencar C, Tamburic L, Brauer M. Descriptive epidemiological features of bronchiolitis in a population-based cohort. Pediatrics. 2008 Dec;122(6):1196-203. doi: 10.1542/peds.2007-2231. PMID 19047234
- [Background] Mansbach JM, Emond JA, Camargo CA Jr. Bronchiolitis in US emergency departments 1992 to 2000: epidemiology and practice variation. Pediatr Emerg Care. 2005 Apr;21(4):242-7. doi: 10.1097/01.pec.0000161469.19841.86. PMID 15824683
- [Background] Jartti T, Jartti L, Ruuskanen O, Soderlund-Venermo M. New respiratory viral infections. Curr Opin Pulm Med. 2012 May;18(3):271-8. doi: 10.1097/MCP.0b013e328351f8d4. PMID 22366993
- [Background] Corneli HM, Zorc JJ, Mahajan P, Shaw KN, Holubkov R, Reeves SD, Ruddy RM, Malik B, Nelson KA, Bregstein JS, Brown KM, Denenberg MN, Lillis KA, Cimpello LB, Tsung JW, Borgialli DA, Baskin MN, Teshome G, Goldstein MA, Monroe D, Dean JM, Kuppermann N; Bronchiolitis Study Group of the Pediatric Emergency Care Applied Research Network (PECARN). A multicenter, randomized, controlled trial of dexamethasone for bronchiolitis. N Engl J Med. 2007 Jul 26;357(4):331-9. doi: 10.1056/NEJMoa071255. PMID 17652648
- [Result] Liu L, Johnson HL, Cousens S, Perin J, Scott S, Lawn JE, Rudan I, Campbell H, Cibulskis R, Li M, Mathers C, Black RE; Child Health Epidemiology Reference Group of WHO and UNICEF. Global, regional, and national causes of child mortality: an updated systematic analysis for 2010 with time trends since 2000. Lancet. 2012 Jun 9;379(9832):2151-61. doi: 10.1016/S0140-6736(12)60560-1. Epub 2012 May 11. PMID 22579125
- [Result] Cantón SBF, Trujillo GG, Uribe RV. Principales causas de mortalidad infantil en México: tendencias recientes. Bol Med Hosp Infant Mex. 2012;69(2):144-8.
- [Result] Cincinnati Children's Hospital Medical Center. Evidence-based care guideline for management of first time episode bronchiolitis in infants less than 1 year of age.